CLINICAL TRIAL: NCT06909682
Title: Smart Monitoring and Analysis System Based on Artificial Intelligence for Patients With Chronic Heart Failure Using Advanced Mini-Invasive and Wearable Medical Devices
Brief Title: AI-Based Monitoring System for Chronic Heart Failure With Advanced Wearable and Mini-Invasive Devices
Acronym: SMART-CARE
Status: Not yet recruiting | Type: Observational
Sponsor: University of Salerno (Other)
Responsible Party: Principal Investigator, Alessia Bramanti, Associate Professor, University of Salerno
Other Study IDs: D43C22002120006
Record Dates: First submitted 2025-03-14; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Chronic Heart Failure; Cardiovascular Diseases; Heart Failure With Reduced Ejection Fraction (HFrEF); Heart Failure With Preserved Ejection Fraction (HFPEF); Congestive Heart Failure Chronic
Keywords: Wearable Medical Devices; Remote Patient Monitoring; Artificial Intelligence in Cardiology; Smart Wearables for Healthcare; Observational Study in Heart Failure; AI-Based Predictive Modeling; Telemedicine in Heart Failure; Non-Invasive Health Monitoring; Personalized Medicine for CHF; Quality of Life Improvement in Heart Failure; Heart Failure Readmission Prevention; Telehealth in Chronic Disease Management; Digital Health Solutions for Heart Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The SMART-CARE study will collect and retain the following biospecimens from participants for clinical and research purposes:
  Types of Samples Retained:
  Blood Samples
  * Plasma and Serum - For analysis of biochemical markers related to chronic heart failure (e.g., BNP, NT-proBNP, creatinine, electrolytes, glucose, lipid profile).
  * Urine Samples - To assess kidney function and electrolyte balance. All biospecimens will be pseudo-anonymized and stored securely following ethical guidelines (EU GDPR 2016/679) and institutional biobank policies. Participants will provide specific informed consent for sample retention and potential future res
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Intervention Group (Device Group - AI-Based Remote Monitoring): Participants in this group will wear the EmbracePlus mini-invasive device for continuous remote monitoring over a six-month period. The device tracks key physiological parameters, including oxygen saturation (SpO₂), heart rate variability (HRV), electrodermal activity (EDA), temperature, respiratory rate, and sleep quality. Data is transmitted to a centralized AI-driven platform, which analyzes trends and detects early signs of heart failure worsening. If significant abnormalities are identified, the system triggers automated alerts, prompting teleconsultations or in-person evaluations as needed to ensure timely clinical intervention.
  Interventions: Device: Intervention Group (Device Group - AI-Based Remote Monitoring)
- Control Group (Non-Device Group - Standard Clinical Follow-Up): Participants in this group will receive standard chronic heart failure (CHF) management according to current clinical guidelines. Their follow-up will consist of scheduled in-person visits every three months, during which they will undergo routine laboratory tests (including BNP, NT-proBNP, renal function, and electrolytes), as well as echocardiography and ECG evaluations. Treatment adjustments will be made based on clinical assessments and reported symptoms.
  Interventions: Other: Standard Clinical Follow-Up

INTERVENTIONS:
Device: Intervention Group (Device Group - AI-Based Remote Monitoring) — This intervention utilizes a mini-invasive wearable device for continuous remote monitoring of chronic heart failure (CHF) patients. Unlike traditional telemonitoring, it integrates AI-driven predictive analytics to track oxygen saturation (SpO₂), heart rate variability (HRV), electrodermal activity (EDA), temperature, respiratory rate, and sleep quality in real time. The system generates automated alerts for healthcare providers, enabling early detection of CHF exacerbation and proactive intervention through teleconsultations, medication adjustments, or in-person evaluations. Data is securely transmitted to a cloud-based platform, allowing continuous risk assessment and personalized care adjustments. This approach aims to reduce unnecessary hospitalizations, enhance patient monitoring, and optimize heart failure management through advanced AI-based digital health technology.
  Groups: Intervention Group (Device Group - AI-Based Remote Monitoring)
Other: Standard Clinical Follow-Up — Participants in this group will receive standard chronic heart failure (CHF) management according to current clinical guidelines. Their follow-up will consist of scheduled in-person visits every three months, during which they will undergo routine laboratory tests (including BNP, NT-proBNP, renal function, and electrolytes), as well as echocardiography and ECG evaluations. Treatment adjustments will be made based on clinical assessments and reported symptoms. Unlike the intervention group, these participants will not use a wearable device, and their condition will be monitored exclusively through traditional hospital visits and self-reported health status.
  Groups: Control Group (Non-Device Group - Standard Clinical Follow-Up)

SUMMARY:
The goal of this observational, multicenter study is to evaluate whether AI-driven remote monitoring using a mini-invasive wearable device can improve clinical outcomes in adult patients (≥18 years) with chronic heart failure (CHF).

The main questions it aims to answer are:

* Can continuous remote monitoring reduce hospital admissions (emergency visits and hospitalizations) by 20% compared to standard care?
* Does wearable-based remote monitoring improve functional, biochemical, and instrumental parameters in CHF patients? Researchers will compare patients using the wearable device (intervention group) to those receiving standard clinical follow-up (control group) to assess whether AI-driven monitoring leads to fewer hospitalizations, better disease management, and improved quality of life.

Participants will:

* Wear the EmbracePlus (Empatica Inc.) device continuously for six months (intervention group only).
* Have their biometric data (SpO₂, HRV, EDA, respiratory rate, temperature, sleep quality) monitored remotely.
* Receive automated alerts and teleconsultations if abnormal physiological changes are detected.
* Attend scheduled follow-up visits (remote and in-person) for clinical evaluation and treatment adjustments.

The study aims to provide real-world evidence on whether integrating wearable health technology with AI analytics can enhance CHF management and improve patient outcomes.

DETAILED DESCRIPTION:
Chronic Heart Failure (CHF) is a multifactorial syndrome characterized by high rates of hospitalization, morbidity, and mortality. Despite advances in pharmacological and device-based therapies, early identification of clinical deterioration remains a major challenge. Traditional follow-up models, based primarily on intermittent in-person evaluations, are often inadequate in capturing subclinical changes that precede acute decompensation.

The SMART-CARE (System of Monitoring and Analysis based on Artificial Intelligence for Chronic Heart Failure Patients with Mini-Invasive and Wearable Medical Devices) study aims to assess whether continuous remote monitoring using a CE (Conformité Européenne)-certified wearable device (EmbracePlus by Empatica Inc.) integrated with AI (Artificial Intelligence) analytics can improve the management of CHF patients. The study adopts a prospective, multicenter, observational design with two parallel cohorts: patients managed with standard care versus patients equipped with the wearable device for six months.

The wearable device captures a range of physiological signals-including peripheral capillary oxygen saturation (SpO₂), heart rate variability (HRV), electrodermal activity (EDA), skin conductance level (SCL), respiratory rate, peripheral skin temperature, pulse rate, fatigue detection, and sleep metrics via actigraphy-and transmits them in real time to a centralized digital platform. AI algorithms analyze these data continuously, triggering alerts in the event of abnormal trends. When alerts are generated, patients undergo teleconsultation, with possible treatment adjustments or in-person follow-up as clinically indicated.

The study is designed to generate real-world evidence on whether AI-enhanced monitoring can reduce unplanned hospital admissions by at least 20% over a six-month follow-up, compared to standard care. Secondary endpoints include improvements in cardiac function (evaluated through echocardiographic parameters), neurohormonal biomarkers such as B-type Natriuretic Peptide (BNP) and Atrial Natriuretic Peptide (ANP), exercise tolerance assessed by the Six-Minute Walk Test (6MWT), quality of life measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ), and incidence of therapy-related adverse events (e.g., hypotension, bradyarrhythmias).

In addition to evaluating clinical efficacy, the study supports the development of a predictive multimarker model. Data collected through the SMART-CARE platform-including clinical history, biochemical markers, imaging data, and continuous sensor-derived variables-will be used by collaborating academic centers to train AI algorithms capable of forecasting CHF progression and tailoring individualized interventions.

All data are pseudonymized in compliance with the General Data Protection Regulation (GDPR, Regulation EU 2016/679). The study does not interfere with ongoing medical treatments and adheres to Good Clinical Practice (GCP) and the ethical principles of the Declaration of Helsinki. Patients provide written informed consent prior to enrollment.

The SMART-CARE initiative reflects a broader goal: integrating telemedicine, wearable health technology, and AI-based predictive modeling into a seamless care pathway that promotes proactive CHF management and enables personalized, data-driven therapeutic decisions.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years (adults of any sex)
* Confirmed diagnosis of chronic heart failure (CHF) for at least 6 months prior to screening
* Stable on optimized heart failure therapy for at least one month before enrollment
* Any left ventricular ejection fraction (LVEF) classification, including:

  * Heart Failure with Reduced Ejection Fraction (HFrEF)
  * Heart Failure with Mid-Range Ejection Fraction (HFmrEF)
  * Heart Failure with Preserved Ejection Fraction (HFpEF)
* NYHA Functional Class I, II, or III
* History of at least one hospital admission or outpatient visit in the past 12 months requiring intravenous (IV) diuretics, vasodilators, or inotropes for CHF exacerbation
* Ability to provide written informed consent or availability of a legally authorized representative Exclusion Criteria
* NYHA Functional Class IV or anticipated heart transplant or ventricular assist device (VAD) implantation within 6 months of screening
* Severe renal impairment (eGFR < 30 mL/min/1.73 m²) or dialysis dependence
* Terminal comorbidities (e.g., advanced cancer, end-stage pulmonary disease) significantly limiting life expectancy
* Pregnancy
* Presence of skin conditions or allergies preventing prolonged use of a wearable device
* Inability to comply with study procedures (e.g., cognitive impairment, significant psychiatric disorders)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The SMART-CARE study will enroll adult patients (≥18 years) with chronic heart failure (CHF) from specialized cardiology and geriatrics clinics. Participants will have NYHA Class I-III heart failure and varying left ventricular ejection fraction (LVEF) classifications (HFrEF, HFmrEF, HFpEF).
  Patients will be recruited from tertiary hospitals and research centers, including:
  AOU "San Giovanni di Dio Ruggi d'Aragona" (Cardiology & Cardiac Rehab) IRCCS Neurolesi "Bonino Pulejo" (Cardiology Unit) IRCCS Fondazione Casa Sollievo della Sofferenza (Geriatrics Unit)
  The study will compare:
  Intervention Group: AI-based remote monitoring with a wearable device. Control Group: Standard CHF management with routine follow-ups. Participants will be clinically stable but at risk of hospitalization, and those with NYHA Class IV, severe renal impairment, or terminal illnesses will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Change in Hospital Admissions with AI-Based Remote Monitoring | 6 months from participant enrollment.
  The study aims to determine whether AI-based remote monitoring using a wearable device leads to a 20% reduction in hospital admissions (including emergency department visits and hospitalizations) compared to standard clinical follow-up in patients with chronic heart failure (CHF). The intervention group will use a mini-invasive wearable device for continuous physiological monitoring, while the control group will receive standard CHF management without remote monitoring. Hospital admission rates will be analyzed to assess the effectiveness of early AI-driven detection and intervention.

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline, 3 months, and 6 months
  Quality of life (QoL) will be measured using the Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score, a validated instrument specifically designed to assess symptom burden, functional status, social limitations, and quality of life in patients with chronic heart failure (CHF). The score ranges from 0 to 100, where higher scores indicate better health status and quality of life. The study will evaluate whether patients in the AI-based remote monitoring group report higher KCCQ scores compared to the control group.
  Unit of Measure: KCCQ score (0-100 scale) Time Frame: Baseline, 3 months, and 6 months Interpretation: Higher scores indicate better outcomes.
Adverse Effects of CHF Therapy | 6 months
  The study will analyze whether continuous AI-driven monitoring helps in reducing adverse effects related to CHF treatments, such as:
  Hypotension (low blood pressure episodes due to overuse of diuretics or vasodilators) Bradyarrhythmias (slow heart rate linked to beta-blockers or other heart failure medications) By detecting early physiological changes, the wearable device may enable timely adjustments in medication dosages, reducing complications and therapy-related hospitalizations.
Change in Biochemical Parameters | 3 and 6 months from participant enrollment
  Biochemical Parameters:
  Change in B-type Natriuretic Peptide (BNP) Levels (picograms per milliliter)
Change in Biochemical Parameters | 3 and 6 months from participant enrollment
  Biochemical Parameters:
  Change in N-terminal pro-BNP (NT-proBNP) Levels (picograms per milliliter)
Change in Biochemical Parameters | 3 and 6 months from participant enrollment
  Biochemical Parameters:
  Change in Serum Creatinine (milligrams per deciliter)
Change in Biochemical Parameters | 3 and 6 months from participant enrollment
  Biochemical Parameters:
  Change in Estimated Glomerular Filtration Rate (eGFR) (milliliters per minute per 1.73 square meters)
Change in Biochemical Parameters | 3 and 6 months from participant enrollment
  Biochemical Parameters:
  Change in Serum Sodium Levels (millimoles per liter)
Change in Biochemical Parameters | 3 and 6 months from participant enrollment
  Biochemical Parameters:
  Change in Serum Potassium Levels (millimoles per liter)
Change in Biochemical Parameters | 3 and 6 months from participant enrollment
  Biochemical Parameters:
  Change in Serum Chloride Levels (millimoles per liter)
Change in Functional ECG-Derived Parameters | 3 and 6 months from participant enrollment
  ECG-Derived Parameters:
  Change in Heart Rate Variability (HRV) (milliseconds)
Change in Functional ECG-Derived Parameters | 3 and 6 months from participant enrollment
  ECG-Derived Parameters:
  Change in Respiratory Rate (breaths per minute)
Change in Functional Echocardiographic derived Parameters | 3 and 6 months from participant enrollment
  Echocardiographic Parameters:
  Change in Left Ventricular Ejection Fraction (LVEF) (percent)
Change in Functional Echocardiographic derived Parameters | 3 and 6 months from participant enrollment
  Echocardiographic Parameters:
  Change in Diastolic Function - E/A Ratio (unitless)
Change in Functional Echocardiographic derived Parameters | 3 and 6 months from participant enrollment
  Echocardiographic Parameters:
  Change in Left Ventricular End-Diastolic Volume (milliliters)
Change in Functional Echocardiographic derived Parameters | 3 and 6 months from participant enrollment
  Echocardiographic Parameters:
  Change in Left Ventricular End-Systolic Volume (milliliters)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang WH, Francis GS, Morrow DA, Newby LK, Cannon CP, Jesse RL, Storrow AB, Christenson RH, Apple FS, Ravkilde J, Wu AH; National Academy of Clinical Biochemistry Laboratory Medicine. National Academy of Clinical Biochemistry Laboratory Medicine practice guidelines: Clinical utilization of cardiac biomarker testing in heart failure. Circulation. 2007 Jul 31;116(5):e99-109. doi: 10.1161/CIRCULATIONAHA.107.185267. Epub 2007 Jul 14. No abstract available. PMID 17630410
- [Background] Cleland JG, Daubert JC, Erdmann E, Freemantle N, Gras D, Kappenberger L, Tavazzi L; Cardiac Resynchronization-Heart Failure (CARE-HF) Study Investigators. The effect of cardiac resynchronization on morbidity and mortality in heart failure. N Engl J Med. 2005 Apr 14;352(15):1539-49. doi: 10.1056/NEJMoa050496. Epub 2005 Mar 7. PMID 15753115
- [Background] Bousquet J, Anto JM, Sterk PJ, Adcock IM, Chung KF, Roca J, Agusti A, Brightling C, Cambon-Thomsen A, Cesario A, Abdelhak S, Antonarakis SE, Avignon A, Ballabio A, Baraldi E, Baranov A, Bieber T, Bockaert J, Brahmachari S, Brambilla C, Bringer J, Dauzat M, Ernberg I, Fabbri L, Froguel P, Galas D, Gojobori T, Hunter P, Jorgensen C, Kauffmann F, Kourilsky P, Kowalski ML, Lancet D, Pen CL, Mallet J, Mayosi B, Mercier J, Metspalu A, Nadeau JH, Ninot G, Noble D, Ozturk M, Palkonen S, Prefaut C, Rabe K, Renard E, Roberts RG, Samolinski B, Schunemann HJ, Simon HU, Soares MB, Superti-Furga G, Tegner J, Verjovski-Almeida S, Wellstead P, Wolkenhauer O, Wouters E, Balling R, Brookes AJ, Charron D, Pison C, Chen Z, Hood L, Auffray C. Systems medicine and integrated care to combat chronic noncommunicable diseases. Genome Med. 2011 Jul 6;3(7):43. doi: 10.1186/gm259. PMID 21745417
- [Background] Keijser W, de Manuel-Keenoy E, d'Angelantonio M, Stafylas P, Hobson P, Apuzzo G, Hurtado M, Oates J, Bousquet J, Senn A. DG Connect Funded Projects on Information and Communication Technologies (ICT) for Old Age People: Beyond Silos, CareWell and SmartCare. J Nutr Health Aging. 2016;20(10):1024-1033. doi: 10.1007/s12603-016-0804-0. PMID 27925142
- [Derived] Ciccarelli M, Bramanti A, Carrizzo A, Garofano M, Visco V, Izzo C, Rusciano MR, Galasso G, Loria F, Bruno G, Vecchione C. Artificial intelligence-based remote monitoring for chronic heart failure: design and rationale of the SMART-CARE study. Front Digit Health. 2025 Dec 10;7:1719562. doi: 10.3389/fdgth.2025.1719562. eCollection 2025. PMID 41451381